CLINICAL TRIAL: NCT06905002
Title: Enhancing the Patient Journey to Clinical Trial Enrolment with Navigation to Optimize Accrual: a Pilot Study for a Prospective, Pragmatic Multi-centre, Stepped Wedge, Cluster Randomized Controlled Trial
Brief Title: Enhancing the Patient Journey to Clinical Trial Enrolment with Navigation to Optimize Accrual
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Windsor Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Health Services Research
Other Study IDs: 22-439
Record Dates: First submitted 2025-03-17; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Clinical trials navigator
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Pilot Stepped-Wedge Cluster- Randomized Control Trial
Who Masked: Participant, Care Provider
Masking Description: Patient information will be masked by replacing clinical sensitive information with unique identifiers. Health care professional identifying information will be replaced with unique identifiers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: Patients: Pre and post intervention (Active Comparator): In the two time periods: pre - intervention and post-intervention, patient charts will be reviewed to assess referral to and accrual onto clinical trials outside of their home cancer treatment centre.
  Interventions: Behavioral: Educational program
- Cohort 3: Physicians and Health Care Professionals (Active Comparator): This group will be followed throughout the pre and post intervention period with regular surveys requesting input on number of patients referred to and accrued onto clinical trials outside of the patient's home cancer treatment centre.
  Interventions: Behavioral: Educational program

INTERVENTIONS:
Behavioral: Educational program — Unique educational program that educates health care professionals on the unique advantages of the Clinical Trials Navigator program. This program is reserved for those centres entering the study. An interactive component of the study is central.

SUMMARY:
Less than 5% of patient enter clinical trials, despite the fact that many patients facing cancer are recommended to seek out clinical trials. One challenge of finding a clinical trial, is the lack of clinical trials at the patient's home cancer centre. The Clinical Trials Navigator (CTN) program was established to help patients, their families and heath care providers navigate the clinical trials systems across Canada in order to identify meaningful clinical trials for patients and help them enter those trials.

The CTN program was piloted in Windsor, Ontario and increased clinical trials accrual for this population by 8%. This study plans to roll out to twenty centres across Canada, mimicing the process. This implementation of the CTN program will be tested by adding centres in a sequential fashion until all centres are added over the 12 month period.

The objectives are improved patient enrollment which will be measured by embedded CTNs in each cancer centre, and reporting to the central site.

Pre- and post-implementation structured interviews with administrators, physicians, patients and allied health care professionals will be used to assess uptake of the CTN program in each centre and reveal potential barriers to successful implementation of a nation-wide CTN program.

The ability of the current CTN program to upscale to twenty centres will be measured by turn-around times of patient reports and through the structured interviews.

DETAILED DESCRIPTION:
PROTOCOL SYNOPSIS In Canada, less than 5% of people living with cancer enroll in clinical trials. The rate of enrollment in trials is even lower among rural populations. The most common barrier to trial enrollment, impacting 30 - 60% of individuals living with cancer, is lack of availability of clinical trials (1-3).

To address this barrier, the Clinical Trials Navigator (CTN) program was developed with support from the Canadian Cancer Clinical Trials Network (3CTN)(4, 5) and hosted by the Windsor Regional Hospital (WRH) in 2019. The objective of this CTN Pilot Trial is to determine the the effectiveness of the CTN program in increasing trial referral rates in twenty new centers across Canada. If we demonstrate that the CTN program can increase the rate of referral to trials across diverse sites in Canada, the CTN program will be a viable solution to overcoming one of the most significant barriers to trial enrollment, thereby advancing treatments and improving outcomes for people living with cancer.

1. THE NEED FOR A TRIAL 1.1.1 What is the problem to be addressed? Clinical trials remain the gold standard to advancing treatments and improving outcomes for people living with cancer. Less than 5% of people living with cancer enroll in trials. The rate of trial enrollment is even lower in rural populations and community hospitals, which account for 65% of hospitals in Canada.(1-3). The most common barrier to trial enrollment, impacting 30 - 60% of individuals living with cancer, is lack of availability of clinical trials, especially among those treated in smaller centres(1-3). Trial availability in Canada ranges from one to 350 trials per center, with larger urban academic centers having more available trials. [Appendix A Accrual by site]. This means many people living with cancer in Canada will be referred to trials that are not available in the center where they receive the majority of their cancer treatment (i.e., a patient's treating cancer center). Stakeholders agree the process of identifying available trials outside of a patient's treating cancer center is the most important barrier currently preventing trial accrual in Canada. (6, 7). 1.1.2 The Clinical Trials Navigator (CTN) Program Structure In 2019, the CTN program was designed in collaboration with key stakeholders, including with people with lived experience (PWLE), to resolve the gap in navigating enrollment into available trials. The CTN program currently incorporates several key components to enhance the trial enrollment process: (i) Publicly accessible referral process through the 3CTN website and posters in the WRH [Appendix B url] [Appendix C poster] (ii) Expert navigators trained in conducting thorough searches to identify available trials (iii) Continuous quality improvement through tracking key metrics that inform ongoing optimization of the CTN program (iv) Knowledge dissemination including sharing best practices and valuable insights with the broader community.

   1.1.3 The Effectiveness of the CTN Program The process from initial referral to the CTN program to trial enrollment is outlined in Appendix D.

   Since inception in 2019, over 600 patients from across Canada have been referred to the CTN program, with 26% being referred to a clinical trial and 8% enrolling in an interventional clinical trial (8). An ongoing iterative process allowed the following improvements: (i) a new EDI survey which allowed users to self-identify as evidenced by one aboriginal and one trans-gender person in our database, (ii) Master Lists for all major cancer types have been developed to overcome challenges of search engines (7). We have demonstrated these master lists increase meaningful trial identification over existing resources [Appendix E, Master List]

   1.1.4 Ongoing CTN program optimization The need to continue to scale the CTN program across Canada is evidenced by the fact that 75% of patients using the CTN program are from the host site. The following objectives were developed by the CTN program Steering Committee for this grant: (i) increase engagement of PWLE and healthcare professionals with the CTN program, (ii) clarify trial eligibility criteria, and (iii) ensure ability of the CTN program to up-scale to increasing demand. 1.2 What is the principal research question to be addressed? Does this pilot multi-center, stepped wedge, cluster randomized controlled trial (SW-RCT) trial assessing the effectiveness of the CTN program demonstrate an increase in clinical trial referral rates? 1.3 Why is the trial needed now? Current initiatives to address poor clinical trials accrual include CRAFT(9), ACRO(10) and CATCH-UP.2020(10). CRAFT and ACRO focus on decentralizing clinical trials, bringing clinical trials to remote patients. CATCH-UP.2020, a NIH supported initiative, focuses on accruing a more diverse population and they have identified navigators as one of the most effective processes to increase accrual to trials. Marathon of Hope (MoH) Cancer Centres in Canada(11) focuses on expanding access for Canadian patients to full genomic profiling. CTN is complementary to these initiatives as has been acknowledged by MoH and 3CTN. In addition, the Canadian Cancer Trials website(12) previously sponsored by the Canadian Cancer Society was sunsetted in July 2023 leaving a gap in service to Canadian patients that can be supported by the CTN program.

   1.4 How will the results of this trial be used? The results of this successful, SW-RCT will establish the CTN program as a vital component of a successful clinical trials ecosystem in Canada. 1.4.1 Knowledge translation We will leverage our association with the patient advocacy groups (e.g., Save Your Skin and My Gut Feeling), 3CTN, Q-CROC and MoH. Key knowledge translation activities include formal presentation of results to knowledge users and researchers at local, national and international scientific meetings dissemination and of results to patients, healthcare providers and the general public through the online resources of our collaborators as well as publication in open-access medical journals. 1.5 Are there any risks to the safety of participants in the trial? It is estimated that only 50% of patients will identify an available trial for which they are eligible and only 8% of patients will actually enroll in available trials. The CTN program may inadvertently create unrealistic hopes among patients regarding the availability and efficacy of trials. We will provide clear and realistic information during the informed consent process.
2. THE PROPOSED TRIAL 2.1 What is the proposed trial design? This multi-center SW-RCT comparing current standard of care processes for navigating the process of enrollment in clinical trials to the CTN program. 2.2 What are the planned trial interventions? Both experimental and control. In the control arm, centers will continue with their standard-of-care process for identifying available trials and enrollment without direct intervention from the CTN program. In the 2

   treatment arm, people living with cancer and healthcare professionals will be able to use the CTN program to navigate the process for identifying available trials and enrollment.

   2.3 What are the proposed practical arrangements for allocating participants to trial groups? In this trial, two participating centres will enter the trial using their current standard of care for navigating the process of enrollment in clinical trials (i.e., 'standard-of-care period') in this stepped- wedge, cluster randomized controlled trial (SW-RCT). After three months, the CTN program will be implemented at the second centre. To prevent any contamination, a washout period of one month will occur after the CTN program is first implemented at each centre to provide an opportunity to resolve any local issues or challenges that may arise during implementation of the CTN program. The primary comparison will be the post-implementation period, comparing it to the standard- of-care period. Figure 1: Timeline for the trial activities (Blue represents standard-of-care period and yellow represents post-implementation period)

   2.4 What are the proposed methods for protecting against sources of bias? Blinding will not be possible with this intervention by the nature of the study. Allocation to use of CTN team will occur at each site over 12 months, consistent with the stepped wedge design, selected by the study statistician. 2.5 What are the planned inclusion/exclusion criteria? Two pilot centers were selected based on the cluster inclusion criteria, namely representation of diverse settings and populations across Canada and willingness and capacity to participate actively in the pilot study activities. Individual participant inclusion criteria is pragmatic and inclusive. Any physician at a participating center involved in the care of patients with breast cancer will be included. Consenting patients (or their legal guardians for those less than 18 years of age or older) receiving treatment for breast cancer at a participating center will also be eligible to participate in the study. .

   2.6 What is the proposed duration of treatment? The entire study will last 12 months. All sites will participate throughout this period. Using the SW-RCT design, centres will have varied exposure to the CTN program. It is expected that the CTN program will become a permanent program within each of these centers after completion of the trial.

   2.7 What is the proposed frequency and duration of follow up? Physician surveys and stakeholder interviews will occur. There is no follow-up beyond the end of the 12-month study period. Monthly surveys will be distributed through REDCap to all eligible physicians at participating centers to collect information on the numbers of reported patients referred to and enrolled onto clinical trials. Interviews will be held before and after the intervention of the CTN program regarding their attitudes toward the CTN program, including administrative, patient and physician challenges with referral to the CTN program and available trials. 2.8 What are the proposed primary and secondary outcomes? The primary outcome is the referral rate of patients by their treating oncologist to available trials identified through the CTN program. This is defined as the number of patients who have clinical trials referral divided by the number of patients seen at each site having metastatic breast malignancy during the study period. The key secondary outcomes include clinical trial accrual rate, stakeholder attitudes towards the CTN program, barriers to clinical trial referral and enrollment and the ability of the CTN program to upscale to increased demands. 2.9 How will the outcomes measures be measured at follow-up? The primary and secondary outcomes will be measured by an embedded 0.2 FTE at each site identifying clinical trials referral to trials outside of the home site, through monthly physician surveys (physician-reported patient referred and enrolled) and structured stakeholder interviews as per Figure 1. Turnaround times for stakeholder reports for stakeholder from the CTN program will be maintained to assess scalability of the CTN program to increase demand as a result of the pilot trial.

   2.10 Proposed sample size At each of the two sites, it is estimated that 60 new patients with the selected cancers are seen each month. It is also estimated that currently, 3% of patients get referred, while use of a CTN team can increase this number to approximately 26% (based on current results observed at the Windsor site).

   Based on these assumptions, a one-sided, alpha=0.10 stepped wedge cluster randomized test with intra- class correlation of 0.001, would have in excess of 82% power to detect a difference. Power calculations are based on the WaldZ-test (calculated using NCSS PASS version 22.0.3). 2.11 Are health services research issues addressed? Clinical trials accrual is a persistent and serious problem in health care delivery. Poor accrual increases costs to the entire health care system, delaying and increasing costs of the discovery of new therapies. If the CTN program is successful at improving trial accrual, it will directly address this health services issue. We have also partnered with Save Your Skin Foundation to learn their process for minimizing financial, policy and social barriers to trial enrollment. 2.12 Planned recruitment rate? How will the recruitment be organized? Over what time period? What evidence that this is achievable. Based on the experiences of implementing the CTN program at WRH, it is anticipated that the CTN Program will be fully implemented within the required timeframe for trial activities. The estimated number of patients with metastatic breast, melanoma, sarcoma and gastrointestinal cancer are estimated based on population data and are a conservative estimate to ensure a realistic recruitment rate.

   2.13 Are there likely to be challenges with compliance? A variation in referral to the CTN program is expected, with thirteen of the fifteen oncologists at the initial WRH site providing a median of 7 referrals per physician per year (range of 1 - 21 referrals per physician). We have increased the implementation activities with this pilot study and anticipate a higher rate of referrals to the CTN program as a result. 2.14 What is the likely rate of loss of follow-up? No patient should be lost to follow-up in this design, as we will engage a part-time research associate at each site with access to patient charts to ensure complete follow-up. 2.15 How many centres will be involved? Two centres will be included in this study. Summary statistics will be used to describe patient and physician characteristics, as well as outcomes of interest. We will compare the number of patients referred pre- and post-intervention using a repeated measures generalized linear regression model. Results will be presented along with 95% confidence intervals. All analyses other than the primary outcome analysis will be two-sided. 2.17 What is the proposed frequency of analyses? Analyses will be conducted at the completion of the trial. There are no planned interim analyses. 2.18 Are there any planned subgroup analyses? The primary objective of the pilot trial is to assess feasibility without subgroup analyses.
3. Trial Management The trial will be coordinated by the established CTN program in Windsor. Dr. Hamm will be the study sponsor. As we currently are available nationally, this will not change the day-to-day management of our program. We will continue to use the REDCap based survey and the data management system with established quality assurance protocols. Statistical analysis will receive oversight by the biostatistician. 3.1 What are the arrangements for day-to-day management of the trial? Who is responsible for coordination? We will continue to use the current processes for the CTN program. The lead navigator is responsible for interaction and engagement with stakeholders, interacting with site CRAs to ensure accurate clinical trials searches, enrollment of patients onto the REDCap database. Dr.

Hamm will hold the primary responsibility for oversight of the program. 3.2 What will be the role of each principal applicant and co-applicant proposed? See Appendix H 3.3 Describe the steering committee and if relevant the data safety monitoring committee.

The steering committee of this program is led by Drs. Hamm and Delisle. The steering committee includes Drs Laferriere, Butler, Perera, Petrella and Greg Pond and Diane Marley. As there is minimal risk to patents, a DSMB is not relevant.

ELIGIBILITY:
Inclusion Criteria:

* Limited to Thunder Bay and Winnipeg health care professionals and patients;

Exclusion Criteria:

* People outside of these two expansion sites

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
At least a 10% increase in the number of patients from Thunder Bay and Winnipeg referred to clinical trials outside of the patient's home cancer treatment site. | 12 months
  Following the intervention, increased awareness of the program will increase the numbers of cancer patients referred to clinical trials at sites outside of the treating site.
At least a 5% increase in the number of patients from Thunder Bay and Winnipeg enrolled onto clinical trials outside of the patient's home cancer treatment site. | 12 months
  Following the intervention, increased awareness of the program will increase the numbers of cancer patients enrolled onto clinical trials at sites outside of the treating site.

SECONDARY OUTCOMES:
Health Care Professional Interviews | 12 months
  Physicians and health care professionals will be interviewed using the CFIR guidelines to obtain potential barriers and opportunities for optimization of the CTN program.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline M Hamm, MD, Principal Investigator — Western Unversity

IPD SHARING:
Plan to Share IPD: Yes
Only aggregate patient data will be used for research presentation, however in order to publish this data, we will share the de-identified patient data in the process of manuscript publication.
Supporting Information: Study Protocol, ICF